CLINICAL TRIAL: NCT01208402
Title: Safety and Efficacy of Esmolol for the Treatment of Peri-operative Tachycardia in Patients at Risk for Post Operative Adverse Ischemic Outcomes
Brief Title: Esmolol for Treatment of Perioperative Tachycardia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Baxter has terminated the study for inadequate enrollment rate accrual.
Sponsor: Duke University (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00024224
Record Dates: First submitted 2010-09-10; First posted 2010-09-24 (Estimated); Results first posted 2014-11-19 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-11

CONDITIONS: High-risk, Non-cardiovascular Surgeries
MeSH Terms: interventions — esmolol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- oral long acting beta blocker (Active Comparator): oral administration of long acting beta blocker as standard of care on the day of surgery
  Interventions: Drug: Esmolol
- Esmolol infusion (Experimental): given 30 minutes prior to induction up to 12 hours post-op
  Interventions: Drug: Esmolol

INTERVENTIONS:
Drug: Esmolol — Infusion will be started at 50 mcg/kg/min for 4 minutes and titrated in increments of 50 mcg/kg/min up to a maximum of 300mcg/kg/min (maintenance dose) to maintain a heart rate between 60 and 80 beats per minute (bpm) while maintaining a minimum systolic blood pressure (SBP) of 95 mmHg during the length of surgery and up to 12 hours post-operatively.
  Other Names: Brevibloc

SUMMARY:
The purpose of this study is to find out if Esmolol is a safe and effective alternative treatment compared to standard treatment using a long acting beta blocker drug, in controlling abnormal heart rate before, during and immediately after surgery.

DETAILED DESCRIPTION:
The benefit versus risk of perioperative beta blockade therapy for adverse ischemic event risk reduction in high risk patients undergoing non-cardiac surgery has been recently challenged. In particular the PeriOperative Ischemia Study Evaluation (POISE trial) showed a cardio-protective effect only at the expense of a higher incidence of stroke and all-cause mortality . In that study death and stroke were significantly associated with an increase in hypotension and bradycardia. Long acting agents - aggressively administered to achieve heart rate (HR) control - appear to be associated with significant adverse outcomes (death, stroke) despite myocardial ischemia and infarction reduction.

It is estimated that 20 percent of high risk patients come to surgery with chronic beta blocker oral therapy. The American Heart Association recommends continuation of beta blockers in this situation as beta-blocker withdrawal is associated with increased rate of perioperative myocardial infarction . Protocols optimizing the perioperative administration of beta-blockers in high-risk patients are therefore needed.

Esmolol is a cardioselective beta-blocker with a short elimination half-life (t1/2 = 9.2 min) and no intrinsic sympathomimetic activity. Evidence has revealed that Esmolol, with its unique short half life can be quickly titrated to both achieve a target hemodynamic effect as well as reduce (or loose) its effect quickly in unstable situations thereby mitigates undesired hypotension and / or bradycardia.

This study proposes to assess the Safety and Efficacy of dosing to target endpoints with Esmolol - an ultra short acting beta blocker - the day of surgery compared to standard long acting oral Metoprolol the day of surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Males or Females
2. Age > 40y/o
3. Scheduled high risk (ASA II-IV) non-cardiac surgery with anticipated 12 hour post-operative ICU care
4. Written informed consent
5. Patients on a stable chronic oral beta-blocker therapy
6. Revised Cardiac Risk Index 1(below) Cardiac Risk Index 1 or greater (below)

   * a history of coronary disease
   * a history of congestive heart failure
   * a history of treated diabetes
   * a history of cerebrovascular disease
   * a history of chronic renal failure

Exclusion Criteria:

1. Active bleeding
2. Untreated left main disease
3. Active cardiac condition (eg unstable angina pectoris, acute exacerbation of CHF, serious arrhythmias, symptomatic valve disease)
4. Preoperative positive troponin T
5. Contraindication for esmolol use
6. Previous allergy or intolerance to esmolol
7. Cancer with an expected life expectancy < 6 months
8. Pregnancy or lactating or planning to become pregnant
9. Failure to provide informed consent, unable to understand or follow instructions.
10. History of drug allergy or idiosyncrasy to beta-adrenergic drugs
11. Recent history (within 1 year) of drug or alcohol abuse
12. Patients with a Pacemaker
13. Abnormal liver function Child-Pugh - B
14. Body Mass Index > 45
15. Reactive airway disease (defined as a history of hospitalization with status asthmaticus within the past one year)
16. Surgery scheduled to begin after 2pm

Min Age: 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2010-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Solomon Aronson, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Durham VA Medical Center, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 76 subject signed consent. 58 subjects met all inclusion/exclusion criteria and were randomized into the study.
Groups:
- Long-Acting Beta Blocker: Administer patient's routine oral long acting beta blocker on day of surgery (standard of care).
- Esmolol: Replace patient's routine oral long-acting beta blocker on day of surgery with a bolus of 500 mcg/kg at start of surgery, followed by a 4 minute infusion at 50 mcg/kg/min, titrating up to a maximum of 300mcg/kg/min to maintain heart rate and SBP within specified thresholds during the length of surgery and continuing through 12 hours post-operatively.
Period: Overall Study
Arm/Group | Long-Acting Beta Blocker | Esmolol
Started | 31 | 28
Completed | 30 | 28
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Long-Acting Beta Blocker | Esmolol | Total
Number analyzed (Participants) | 31 | 28 | 59
Age, Customized [Number; unit: participants]
  18 years and older | 31 | 28 | 59
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 22 | 21 | 43
Region of Enrollment [Number; unit: participants]
  United States | 31 | 28 | 59

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Intraoperative Case Time With Heart Rate (HR) <60 or >80 Bpm
Description: Duration of intraoperative excursion (ie, time spent) outside Target HR range defined as 60 to 80 bpm during surgery, expressed as percent of case minutes. Vital signs are measured from start of surgery to end of surgery at 5 minute intervals or less.
Time Frame: Start of surgery to end of surgery, an average duration of 245 minutes
Population: Three enrolled cases (1 in the oral long acting beta blocker group and 2 in the Esmolol infusion group) were excluded from calculations a priori because they received diltiazem, a calcium channel blocker which lowers heart rate, before the operation.
Measure: Median (Inter-Quartile Range); unit: percentage of case minutes
Arm/Group | Long-Acting Beta Blocker | Esmolol
Number analyzed (Participants) | 30 | 26
percentage of case minutes | 39.2 [13.6 to 83] | 37.3 [14.4 to 64.6]

2. Secondary Outcome: Percentage of Intraoperative Case Time With Systolic Blood Pressure <95 mmHg
Description: Duration of intraoperative case time patient was not in the target window of SBP > 95 mmHg, expressed as percent of total case minutes. SBP is measured from start of surgery to end of surgery at 5 minute intervals or less.
Time Frame: Start of surgery to end of surgery, an average duration of 245 minutes
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of surgery minutes
Arm/Group | Long-Acting Beta Blocker | Esmolol
Number analyzed (Participants) | 30 | 26
percentage of surgery minutes | 3.3 [0 to 9.1] | 3.1 [0 to 9.0]

3. Primary Outcome: Percentage of Postoperative First Three Hours With Heart Rate (HR) <60 or >80 Bpm
Description: Duration of postoperative first three hours spent outside Target HR range defined as 60 to 80 bpm, expressed as percent of the total 3 hours. Vital signs are measured from end of surgery to 3 hours postoperatively at 5 minute intervals for the first hour and every 15 minutes thereafter.
Time Frame: End of surgery to 3 hours
Population: Ten cases (7 in the oral long acting beta blocker group and 3 in the Esmolol infusion group) were missing some of the postoperative vital sign measurements, resulting in gaps too long for valid calculation of the postoperative outcomes only.
Measure: Median (Inter-Quartile Range); unit: percentage of 3 hour interval
Arm/Group | Long-Acting Beta Blocker | Esmolol
Number analyzed (Participants) | 23 | 23
percentage of 3 hour interval | 56.5 [8.0 to 93.8] | 39.2 [8.3 to 79.6]

4. Secondary Outcome: Percentage of Postoperative First Three Hours With Systolic Blood Pressure <95 mmHg
Description: Duration of postoperative first three hours patient was not in the target window of SBP > 95 mmHg, expressed as percent of the total 3 hours. SBP is measured from end of surgery to 3 hours postoperatively at 5 minute intervals for first hour and every 15 minutes thereafter.
Time Frame: end of surgery to 3 hours
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: percentage of 3 hour interval
Arm/Group | Long-Acting Beta Blocker | Esmolol
Number analyzed (Participants) | 23 | 23
percentage of 3 hour interval | 0 [0 to 1.4] | 0 [0 to 6.4]

5. Primary Outcome: Percentage of Postoperative Hours 4 to 12 With Heart Rate (HR) <60 or >80 Bpm.
Description: Duration of postoperative hours 4 to 12 spent outside Target HR range defined as 60 to 80 bpm, expressed as percent of the total 9 hours. Vital signs are measured during hours four and five at 30 minute intervals and once every hour for the next 7 hours, through 12 hours postoperatively.
Time Frame: Postoperative hours 4-12
Population: Specific vital sign measurements were available for calculation of outcomes during the final 9 hours postoperatively in 18 cases in the Long-Acting beta blocker group and in 16 cases in the Esmolol group.
Measure: Median (Inter-Quartile Range); unit: percentage of 8 hour interval
Arm/Group | Long-Acting Beta Blocker | Esmolol
Number analyzed (Participants) | 18 | 16
percentage of 8 hour interval | 39.5 [14.2 to 69.8] | 37 [8.2 to 56.9]

6. Secondary Outcome: Percentage of Postoperative Hours 4 to 12 With Systolic Blood Pressure <95 mmHg
Description: Duration of postoperative hours 4 to 12 patient was not in the target window of SBP > 95 mmHg, expressed as percent of the total 9 hours. SBP was measured during hours four and five at 30 minute intervals and once every hour for the next 7 hours, through 12 hours postoperatively.
Time Frame: Postoperative hours 4-12
Population: Specific vital sign measurements were available for calculation of outcomes during the final 9 hours postoperatively in 18 cases in the Long-Acting BB group and in 16 cases in the Esmolol group.
Measure: Median (Inter-Quartile Range); unit: percentage of 8 hour interval
Arm/Group | Long-Acting Beta Blocker | Esmolol
Number analyzed (Participants) | 18 | 16
percentage of 8 hour interval | 0 [0 to 12.2] | 6.8 [0 to 15.2]

ADVERSE EVENTS:
Arm/Group | Long-Acting Beta Blocker | Esmolol
Serious Adverse Events (participants affected / at risk) | 2/31 | 2/28
Other Adverse Events (participants affected / at risk) | 16/31 | 19/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Long-Acting Beta Blocker (N=31) | Esmolol (N=28)
Intra-abdominal retroperitoneal abscess (Gastrointestinal disorders) | 1 | 0
Change in Mental Status (Psychiatric disorders) | 1 | 0
Hemorrhage (Blood and lymphatic system disorders) | 0 | 1 — Hemorrhage status post aortobifemoral bypass
myocardial infarction (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Long-Acting Beta Blocker (N=31) | Esmolol (N=28)
HYERTENSION (Cardiac disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 0 | 1
HEARTBURN (Gastrointestinal disorders) | 0 | 1
HYPOMAGNESEAMIA (Blood and lymphatic system disorders) | 0 | 1
Low urine output (Renal and urinary disorders) | 1 | 0
Urinary tract infection (Renal and urinary disorders) | 2 | 0
NAUSEA (Gastrointestinal disorders) | 2 | 0
DIARRHIA (Gastrointestinal disorders) | 2 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0
CONFUSION (Nervous system disorders) | 1 | 0
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 | 0
DIFFICULTY OF BREATHING (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DIAPHORESIS (Cardiac disorders) | 0 | 1
ILEUS (Gastrointestinal disorders) | 0 | 3
WOUND INFECTION (Infections and infestations) | 0 | 1
CHEST PAIN (Cardiac disorders) | 1 | 1
TACHYCARDIA (Cardiac disorders) | 4 | 4
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Decrease urine output (Renal and urinary disorders) | 1 | 0
Intra-abdominal retroperitoneal abscess (Infections and infestations) | 1 | 0
Mildly elevated serum creatinine (Renal and urinary disorders) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
Fever (General disorders) | 1 | 0
PULMONARY EDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HYPERNATREMIA (Blood and lymphatic system disorders) | 1 | 0
CHANGED MENTAL STATUS (Nervous system disorders) | 1 | 0
HYPOTENSION (Cardiac disorders) | 4 | 4
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HYPONATREMIA (Blood and lymphatic system disorders) | 1 | 0
HYPOKALEMIA (Blood and lymphatic system disorders) | 1 | 0
DIFUSE BRAIN DISFUNCTION (Nervous system disorders) | 1 | 0
POST-SURGICAL BLEEDING (Surgical and medical procedures) | 0 | 1
POST-SURGICAL HEMATOMA (Surgical and medical procedures) | 0 | 1
ANEMIA (Blood and lymphatic system disorders) | 0 | 1
None reversible ischemia in the inferior right heart (Cardiac disorders) | 1 | 0
Agitation (Nervous system disorders) | 1 | 0
DELIRIUM TREMENS (Nervous system disorders) | 0 | 1
Mild right hydronephrosis (Renal and urinary disorders) | 0 | 1
INTRA-OPERATIVE BLEEDING (Surgical and medical procedures) | 1 | 0
BRADYCARDIA (Cardiac disorders) | 0 | 1
Elevated troponin (Cardiac disorders) | 0 | 3
Heavy feeling bilateral arm (Musculoskeletal and connective tissue disorders) | 1 | 0
Clumsiness left arm (Musculoskeletal and connective tissue disorders) | 1 | 0
Apresthesia (General disorders) | 1 | 0
Significant SQ air with SOB (Respiratory, thoracic and mediastinal disorders) | 1 | 0
POST DISCHAGE PAIN (Surgical and medical procedures) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No